CLINICAL TRIAL: NCT00596349
Title: Quality of Life in Women Surviving Ovarian Cancer
Brief Title: Women Surviving Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Queens Cancer Center of Queens Hospital (Other)
Responsible Party: Martee Hensley, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 04-131
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Epithelial Ovarian Cancer; Quality of Life; Survivorship
Keywords: epithelial Ovarian Cancer; Quality of Life; Survivorship
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- A: epithelial ovarian cancer survivors (women disease-free at 5 to 10 years from diagnosis of ovarian cancer)
  Interventions: Behavioral: questionnaires
- B: women in second- or greater remission (women who have had one or more relapses from ovarian cancer but are considered to be currently clinically disease-free 5 to 10 years from original diagnosis of ovarian cancer).
  Interventions: Behavioral: questionnaires
- C: women surviving with epithelial ovarian cancer (women alive with disease 5 to 10 years from original diagnosis of ovarian cancer)
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — study participants complete one-time survey, questionnaires, and cognition testing, comprising the following: QOL-Cancer Survivor FACT-Ovarian SF-36 (general QOL scale) CES-D (depression scale) Impact of Events Scale (anxiety scale) FACT-GOG-NTX (neurotoxicity scale) Female Sexual Functioning Index (FSFI) Cognition Testing Perception of disease chronicity/acuity Concerns about Recurrence Report of surveillance type, frequency, utility Health behaviors Self-report of co-morbidities Self-report of potential unmet needs Background information form List of current medications Patient-defined QoL domains
  Groups: A
Behavioral: questionnaires — study participants complete one-time survey, questionnaires, and cognition testing, comprising the following: QOL-Cancer Survivor FACT-Ovarian SF-36 (general QOL scale) CES-D (depression scale) Impact of Events Scale (anxiety scale) FACT-GOG-NTX (neurotoxicity scale) Female Sexual Functioning Index (FSFI) Cognition Testing Perception of disease chronicity/acuity Concerns about Recurrence Report of surveillance type, frequency, utility Health behaviors Self-report of co-morbidities Self-report of potential unmet needs Background information form List of current medications Patient-defined QoL domains
  Groups: B
Behavioral: questionnaires — study participants complete one-time survey, questionnaires, and cognition testing, comprising the following: QOL- Cancer Survivor, FACT-Ovarian, SF-36, CES-D, IES, FACT-GOG-NTX, FSFI, Cognition Testing, Perception of disease chronicity/acuity, Report of surveillance type, frequency, utility, Health behaviors, Self-report of co-morbidities, Self-report of potential unmet needs, Background information form, List of current medications,Patient-defined QoL domains
  Groups: C

SUMMARY:
The purpose of this study is to help us learn more about how women who have had or now have ovarian cancer are doing 5 years or more from their diagnosis. We want to learn about general quality of life, long-term side effects of treatment, sexual function, thinking, memory, and psychological effects (such as anxiety and depression). We will also look at how these women are being followed for ovarian cancer. We hope this study will help us better understand how women surviving ovarian cancer are doing.

ELIGIBILITY:
Inclusion Criteria:

* Women with invasive epithelial ovarian cancer who are disease-free and 5 to 10 years from diagnosis (for Cohort A) and have never experienced a recurrence of epithelial ovarian cancer
* Women with epithelial ovarian cancer who have had one or more relapses, but are clinically currently disease-free, 5- to 10 years from diagnosis (for Cohort B)
* Women with current evidence of epithelial ovarian cancer who are alive with disease 5 to 10 years from diagnosis (for Cohort C)
* Fluency in English
* Written informed consent

Exclusion Criteria:

* Inability to read, communicate in English
* ovarian cancer of low malignant potential (borderline tumors)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Memorial Sloan-Kettering Cancer Center (MSKCC) clinic The Queens Cancer Center Hospital(QCC)clinic
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2004-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
QOL, phys funct status score on FACT & ,psychol status , cognitive functioning, Brief test of Attention, sexual funct & health behaviors among ovar ca survi & among women in 2nd or > remiss & among women surv with ovar ca 5 to 10 yrs from dx. | conclusion of study

SECONDARY OUTCOMES:
Identify potential determinants of global QOL in all three ovarian cancer survivor cohorts. | conclusion of study

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org